CLINICAL TRIAL: NCT05082532
Title: Efficacy and Safety of Interwoven Self-Expandable Nitinol Stent for Femropopliteal Arterial Occlusive Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Naser Hussein, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUPERA
Record Dates: First submitted 2021-09-03; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Femoropopliteal Occlusive Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with critical and subcritical femoropopliteal arterial occlusions (Experimental): patients presented with chronic ischemia in rest pain stage or ulcerative and gangrenous toes and by investigations long chronic total occlusion of femoropopliteal segment was documented may need stenting of the diseased segment especially if the lesion recoils after previous angioplasty. Nitinol interwoven stent has a unique design that achieves adherence to vessel wall and also malleability with the vessel and surrounding muscle motion so investigators predict more extended patency time with this interventional option and want to investigate this prediction using a scientific experimental pathway.
  Interventions: Other: Interwoven supera stent (IW; Supera Veritas®; Abbott Vascular, Santa Clara, CA, USA) .

INTERVENTIONS:
Other: Interwoven supera stent (IW; Supera Veritas®; Abbott Vascular, Santa Clara, CA, USA) . — we here conduct a prospective study to evaluate the efficacy and safety of self- expandable nitinol stent especially interwoven supera stent (IW; Supera Veritas®; Abbott Vascular, Santa Clara, CA, USA) in femoropoliteal complex occlusive lesions.

SUMMARY:
Interwoven self-expandable stent is a recent endovascular method to treat complex femoropopliteal lesions trying to reach a reasonable patency and durability like in surgical bypass.

DETAILED DESCRIPTION:
Stenting of the femoro-popliteal segment is indicated in case of elastic recoil, flow-limiting dissection, insufficient per- cutaneous transluminal angioplasty (PTA) or long lesion length. However, in-stent restenosis (ISR) or fracture after endovascular treatment remains a serious concern, especially for lesions of a long segment or near the knee joint. Besides the current availability of covered or drug-coated stents, there is the self-expandable bare-metal Nitinol stent which rapidly evolved during the last decade from closed-cell to open-cell and, more recently, to interwoven stents. interwoven nitinol stent design of fully connected structures facilitates a continuous but a traumatic synergy between the stent and vessel wall and hence enables axial compliance. Investigators here conduct a prospective study to evaluate the efficacy and safety of self- expandable nitinol stent especially interwoven supera stent (IW; Supera Veritas®; Abbott Vascular, Santa Clara, CA, USA) in femoropopliteal complex occlusive lesions.

ELIGIBILITY:
Inclusion criteria:

* Patients with critical limb ischemia(grade 4,5&6 Rutherford classification) and patients with disabling claudications which interferes with routine activities (grade 3 Rutherford classification).
* Patients with chronic total occlusion(CTO) of femoropopliteal segment which is equal or beyond 10 centimeters length.
* Patients with recoil after transluminal angioplasty or occlusion in previously deployed stent.
* If the lesion extends to popliteal artey against knee flexion.

Exclusion criteria:

* Pediatric patients.
* Patients with isolated infra-popliteal occlusion.
* Patients with popliteal blind segment with bad runoff.
* Patients with acute thrombotic occlusions.
* Patients with previous bypass surgery in affected limb.
* Patients with aneurysmal lesion in the affected limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
peak systolic velocity in centimeters per second (cm/sec) through the deployed stent in serial duplex imaging | 4 years
  Crossing the lesion and deploying the stent without residual stenosis or degree of stenosis is less than 30% and assess the time the stent remains patent without re interventions. the outcome will be measured on clinical aspect and imaging aspect. Clinically ,investigators will trace the ankle brachial index (ankle systolic pressure relative to systemic systolic pressure), wound healing progress through cascade measuring of ulcer diameter in centimeters till complete healing and pain improvement depending on visual analogue score from 0 to 10.Imaging follow up, investigators will trace diseased segment diameters after intervention in millimeters and peak systolic velocity through the stent in centimeters per second.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mewissen MW. Primary nitinol stenting for femoropopliteal disease. J Endovasc Ther. 2009 Apr;16(2 Suppl 2):II63-81. doi: 10.1583/08-2658.1. PMID 19624075